CLINICAL TRIAL: NCT04561024
Title: Evaluation of a Chest X-Ray AI Neural Network (RadGen SARS-CoV2 Detection System) for the Detection of RT-PCR Confirmed SARS-Cov2 Covid-19 Pneumonia
Brief Title: Evaluation of a COVID-19 Pneumonia CXR AI Detection Algorithm
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ensemble Group Holdings, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: EN-092020
Record Dates: First submitted 2020-09-22; First posted 2020-09-23 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RT-PCR Positive Patients: RT-PCR confirmed patients positive for SARS-CoV-2
  Interventions: Diagnostic Test: AI model
- Negative patients: RT-PCR confirmed patients negative for SARS-CoV-2 or patients with CXR performed before the emergence of COVID-19 pandemic
  Interventions: Diagnostic Test: AI model

INTERVENTIONS:
Diagnostic Test: AI model — Deep Learning CNN model

SUMMARY:
This study investigates the diagnostic performance of an AI algorithm in the detection of COVID-19 pneumonia on chest radiographs.

DETAILED DESCRIPTION:
This is an international multi-center study. Chest radiographs (CXR) from different participating centers will be collected to develop an AI algorithm to detect COVID-19 pneumonia. This will be tested on external hold out datasets from different centers using SARS-CoV-2 by Real-Time Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) Assay as ground truth.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients >18 years of age
* Attended any of the participating institutes between February 1, 2020 until September, 2020
* Underwent both RT-PCR testing and frontal CXR (within 48 hours of PCR testing) for COVID-19 infection
* frontal CXR of patients pre-covid pandemic

Exclusion Criteria:

* Unavailability of patient demographics and clinical data
* Inconclusive RT-PCR results
* CXR considered to be of non-diagnostic quality by the clinical radiology research team at each site
* CXR not in a retrievable or processable format for AI inference

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There will be three subsets of study population in this study; patients who were
  1. RT-PCR confirmed COVID-19 positive
  2. RT-PCR confirmed COVID-19 negative
  3. either had a diagnosis of pneumonia before the 1st January 2020.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance of AI model | 9 months
  Performance (accuracy, sensitivity, specificity, false-positive rate (FPR), false-negative rate (FNR), and Area Under the Curve (AUC)) of the AI model in detection of COVID-19 pneumonia on their baseline CXR using RT-PCR and historical controls as gold standard in a multi-center / multi-national cohort.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No